CLINICAL TRIAL: NCT00579358
Title: Molecular Basis of Congenital Heart Defects
Status: Withdrawn | Type: Observational
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: OCRT07001 [2007-5805]; HS# 2007-5805
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Congenital Heart Defects
Keywords: Congenital heart defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Congenital heart disease is one of the most common malformations in newborns. About 1% of newborns have cardiac malformations. Many need open heart surgery, which contributes substantially to pediatric mortality and morbidity. Recent advances in genetics suggest that many congenital heart defects are caused by mutation of genes. So far, half a dozen genes are found to be associated with congenital heart diseases, such as TBX5, NKX2.5, and GATA4, to name a few. In the near future, more genes will be identified.

This study will evaluate the role of mutation of genes in congenital heart diseases and study the genotype-phenotype correlation. The central hypothesis is that a significant percentage of congenital heart disease is caused by mutation of genes involved in heart development, and the phenotype with missensed mutations is milder than nonsense mutation. Another hypothesis is that a significant proportion of patients with cardiac malformations will have mutations in their genes. The specific aim is to test the mutations of these genes in patients with congenital heart diseases. The study will provide substantial information to understand how the human heart develops. In the future, prenatal diagnosis could be developed based on this study.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to evaluate the role of mutation of genes in congenital heart diseases and study the genotype-phenotype correlation.

Hypothesis:

The central hypothesis is that a significant percentage of congenital heart disease is caused by mutation of genes involved in heart development, and the phenotype with missensed mutations is milder than nonsense mutation. Another hypothesis is that a significant proportion of patients with cardiac malformations will have mutations in their genes. The specific aim is to test the mutations of these genes in patients with congenital heart diseases.

Study Design and Procedures:

This is a pilot study on mutation of genes in congenital heart diseases and genotype-phenotype correlation. Probands and family members are initially evaluated by a local physician or at the UCI Medical Center. A clinical diagnosis is made based on clinical information, echocardiography, EKG, and/or cardiac catheteration.

We would like to correlate the mutation the specific type of congenital heart defect. For example, if mutations of TBX5 more likely cause atrial-septal defects, ventricular-septal defects; mutations PTPN11 is more likely cause pulmonary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children (both parent's signature required) who are able to give informed consent
* Adults or children who are prior diagnosed with congenital heart disease and/or who has immediate family member(s) with congenital heart disease (immediate family members include: subject's parents, siblings, and subject's children)

  * If subject is the only one affected and subject does not disclose of any family member being affected, than only subject will be enrolled
  * If subject is affected and disclose that a family member is affected, that family member will be contacted (with permission) to participate in the study
* Patients of all ethnical origin

Exclusion Criteria:

* Patients diagnosed with no congenital heart disease (as determined by their medical assessment); (if subjects who are unaffected disclose that a family member is affected, with permission, that family will be contacted for participation)
* Patients who are unable to provide informed consent/assent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The characteristics of the proposed subject population include:
  * Children (male or female) who are able to give assent
  * Subjects diagnosed with congenital heart defects
  * Adults (male or female) who are competent to give informed consent
  * Subjects who are unable to read or speak English
  * Individuals of any ethnic origin
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taosheng Huang, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Taosheng Huang, Orange, California, United States